CLINICAL TRIAL: NCT00655928
Title: Modulation of Lung Injury Complicating Lung Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal College of Physicians (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: cro524; 2006-004442-16 (EudraCT Number)
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Acute Lung Injury
Keywords: Acute lung injury; Lung resection
MeSH Terms: conditions — Acute Lung Injury | interventions — Acetylcysteine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): Participant received N-acetylcysteine 240mg/kg in 1 litre 0.9% saline intravenous over 12 hours pre-operatively
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Participant received 0.9% saline 1 litre intravenous over 12 hours pre-operatively
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine 240mg/kg in 1 litre 0.9% saline intravenous over 12 hours pre-operatively
  Arms: N-acetylcysteine
Drug: 0.9% saline — 0.9% saline 1 litre intravenous over 12 hours pre-operatively
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether N-acetylcysteine given intravenously 1 day pre-operatively is effective in preventing inflammation in the lungs, as measured by tests on blood, breath and lung specimens, in patients undergoing surgery to remove a portion of lung.

DETAILED DESCRIPTION:
Acute lung injury occurs following lung resection in about 5% cases, and has a high mortality of around 50%. Management of these patients is largely supportive. Even in patients who do not develop clinical evidence of acute lung injury, markers of inflammation and oxidative stress are present in blood and exhaled breath condensate after lung resection. The purpose of this randomised double-blind placebo-controlled study is to determine whether lung injury can be prevented by pre-administration of N-acetylcysteine.

ELIGIBILITY:
Inclusion Criteria:

* Elective lung resection for cancer

Exclusion Criteria:

* Age less than 18 years
* Women of child-bearing age or potential
* Known allergy to N-acetylcysteine
* Oral steroid in the preceding 1 month
* N-acetylcysteine in the preceding 1 month
* Unable to receive standardised anaesthetic approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Griffiths, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bastin AJ, Davies N, Lim E, Quinlan GJ, Griffiths MJ. Systemic inflammation and oxidative stress post-lung resection: Effect of pretreatment with N-acetylcysteine. Respirology. 2016 Jan;21(1):180-7. doi: 10.1111/resp.12662. Epub 2015 Oct 27. PMID 26503312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine | Placebo
Started | 26 | 26
Completed | 23 | 24
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10.1) | 63.9 (11.5) | 65.95 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 15 | 15 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23 | 24 | 47
Spirometry, FEV1 [Mean (Standard Deviation); unit: litres] | 2.23 (0.97) | 2.56 (0.81) | 2.39 (0.89)
FVC [Mean (Standard Deviation); unit: litres] | 3.48 (1.17) | 3.6 (1.01) | 3.54 (1.09)
Duration of one-lung ventilation [Mean (Standard Deviation); unit: minutes] — One lung ventilation is a process that refers to mechanical separation of the two lungs to allow ventilation of only one lung, while the other lung is compressed by the surgeon or allowed to passively deflate.
  minutes | 134 (42) | 137 (59) | 135.5 (50.5)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Plasma IL-6
Description: Plasma IL-6 was measured in duplicate using ELISA.
Time Frame: Post operative, 24 hours
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 23 | 24
pg/ml | 126 [80 to 180] | 111 [72 to 162]
Statistical Analysis 1: Comparison: N-acetylcysteine vs Placebo; Test type: Superiority; p = 0.09, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | N-acetylcysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 14/23 | 12/24
Other Adverse Events (participants affected / at risk) | 8/23 | 5/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=23) | Placebo (N=24)
Postoperative complication (Surgical and medical procedures) | 13 (13) | 10 (10)
Acut lung injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=23) | Placebo (N=24)
Respiratory infection (Infections and infestations) | 6 (6) | 3 (3)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Pleural fluid infection (Infections and infestations) | 2 (2) | 2 (2)
Intravascular cannula infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The investigator did not sample the pulmonary compartment for markers of inflammation or oxidative damage due to reliance on OLV during surgery, may have led to underestimation of pulmonary inflammation and effect of antioxidant supplementation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes